CLINICAL TRIAL: NCT02817243
Title: The Drug Interaction Study of SP2086 and Simvastatin in Healthy Subjects
Brief Title: The DDI Study of SP2086 and Simvastatin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-112
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP2086 and Simvastatin (Other): SP2086 will be administered orally (by mouth) as 100 mg on Days 4, 5, 6, 7, and 8 and Simvastatin will be administered orally as two 20mg tablets on Days 1 and 8. Both SP2086 and Simvastatin tablets will be taken with 8 ounces (240 mL) of water.
  Interventions: Drug: SP2086; Drug: Simvastatin

INTERVENTIONS:
Drug: SP2086 — SP2086 will be administered orally (by mouth) as 100 mg on Days 4, 5, 6, 7, and 8 and Simvastatin will be administered orally as two 20mg tablets on Days 1 and 8. Both SP2086 and Simvastatin tablets will be taken with 8 ounces (240 mL) of water.
Drug: Simvastatin — SP2086 will be administered orally (by mouth) as 100 mg on Days 4, 5, 6, 7, and 8 and Simvastatin will be administered orally as two 20mg tablets on Days 1 and 8. Both SP2086 and Simvastatin tablets will be taken with 8 ounces (240 mL) of water.

SUMMARY:
The purpose of the study is to investigate the potential interaction between multiple oral doses of SP2086 and a single oral dose of Simvastatin in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center study of SP2086 and Simvastatin in healthy adult volunteers. SP2086 will be administered orally (by mouth) as 100 mg on Days 4, 5, 6, 7, and 8 and Simvastatin will be administered orally as two 20mg tablets on Days 1 and 8. Both SP2086 and Simvastatin tablets will be taken with 8 ounces (240 mL) of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 26 kg/m2

Exclusion Criteria:

* History of diabetes
* History of heart failure or renal insufficiency
* Urinary tract infections, or vulvovaginal mycotic infections
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SP2086 or metformin or any of the excipients of the formulation of SP2086 or Simvastatin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 9
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of Simvastatin.
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 9
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of Simvastatin.
The maximum plasma concentration (Cmax) of Simvastatin | up to Day 9
  Cmax (a measure of the body's exposure to Simvastatin) will be compared. before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 | up to Day 9
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of Simvastatin.
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to Day 9
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of Simvastatin.
The area under the plasma concentration-time curve (AUC) of Simvastatin | up to Day 9
  AUC (a measure of the body's exposure to Simvastatin) will be compared before and after administration of multiple doses of SP2086.

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hosital of Jilin University, Changchun, Jilin, China